CLINICAL TRIAL: NCT02049424
Title: Retrospective-prospective Observational Study for Data Collection of Patients Who Underwent an Haploidentical Transplantation After Non-myeloablative Conditioning Regimen
Brief Title: Observational Study in Patients Who Underwent an Haploidentical Transplantation With T-repleted Bone Marrow
Status: Terminated | Type: Observational
Why Stopped: low recruitment
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: ONC/OSS-03/2011
Record Dates: First submitted 2013-06-28; First posted 2014-01-30 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2014-01

CONDITIONS: Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- transplanted patients: T-repleted haploidentical transplanted patients in Italy

SUMMARY:
Outcome evaluation in patients who underwent transplantation with T-repleted bone marrow after post-transplantation cyclophosphamide

DETAILED DESCRIPTION:
Patients who underwent transplantation with T-repleted bone marrow haploidentical transplantation will be analyzed considering toxicity incidence (GVHD, infective complications, graft-failure incidence and TRM)and efficacy variables (Overall Survival, Progression Free Survival and Relapse incidence)

ELIGIBILITY:
Inclusion Criteria:

- patients affected by hematologic neoplasia who underwent a haploidentical transplantation (2-3 mismatches) from a familiar donor, with non-ex vivo manipulated bone marrow and post-transplantation cyclophosphamide

Exclusion Criteria:

* ex vivo manipulated bone marrow transplantation
* use of antilymphocyte serum during conditioning

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who underwent a haploidentical transplantion after non-myeloablative conditioning regimen
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2011-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
toxicity evaluation | 1 year
  Chronic and acute GVHD, infectious complications, graft failure, TRM

CONTACTS AND LOCATIONS:
Overall Officials: Luca Castagna, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, MI, Italy

REFERENCES:
- [Derived] Roberto A, Castagna L, Zanon V, Bramanti S, Crocchiolo R, McLaren JE, Gandolfi S, Tentorio P, Sarina B, Timofeeva I, Santoro A, Carlo-Stella C, Bruno B, Carniti C, Corradini P, Gostick E, Ladell K, Price DA, Roederer M, Mavilio D, Lugli E. Role of naive-derived T memory stem cells in T-cell reconstitution following allogeneic transplantation. Blood. 2015 Apr 30;125(18):2855-64. doi: 10.1182/blood-2014-11-608406. Epub 2015 Mar 5. PMID 25742699
- [Derived] Roberto A, Castagna L, Gandolfi S, Zanon V, Bramanti S, Sarina B, Crocchiolo R, Todisco E, Carlo-Stella C, Tentorio P, Timofeeva I, Santoro A, Della Bella S, Roederer M, Mavilio D, Lugli E. B-cell reconstitution recapitulates B-cell lymphopoiesis following haploidentical BM transplantation and post-transplant CY. Bone Marrow Transplant. 2015 Feb;50(2):317-9. doi: 10.1038/bmt.2014.266. Epub 2014 Nov 24. No abstract available. PMID 25419693